CLINICAL TRIAL: NCT01723553
Title: Amyloid-related Imaging Abnormalities (Microbleeds) in Atypical AD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jennifer Whitwell, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-007139
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Atypical Alzheimers Disease; Logopenic Variant of Primary Progressive Aphasia (LPA); Posterior Cortical Atrophy (PCA)
Keywords: aphasia; logopenic; PCA; LPA
MeSH Terms: conditions — Aphasia | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PiB positron emission tomography (PET) (Experimental): All subjects will receive PET imaging with C-11 PiB on approximately day 1 or day 2 of study to determine if they have beta-amyloid deposits in their brains.
  Interventions: Drug: C-11 PiB

INTERVENTIONS:
Drug: C-11 PiB — One time intravenous administration of ~740 megabecquerel (MBq) of [N-methyl-C-11]2-(4'-methylaminophenyl)-6-hydroxybenzothiazole (PiB) (range 370 - 740 MBq).
  Other Names: Pittsburgh Compound B; PiB

SUMMARY:
The study is designed to assess the demographic, clinical and imaging associations with the presence of microbleeds in atypical Alzheimer's disease. The primary hypothesis is that cognitive and functional performance will be poorer in atypical Alzheimer's subjects with microbleeds compared to those without microbleeds.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is associated with amyloid-related imaging abnormalities (ARIA). Microbleeds (MBs) represent part of the spectrum of ARIA and can be identified as small hypointense lesions on gradient-recalled echo (GRE) T2*-weighted MRI. They are thought to represent hemosiderin deposits (and hence have been classified as ARIA-H1) and occur as a consequence of leakage of blood products out of vessels that have been damaged by deposition of the protein β-amyloid in cerebral vessels; cerebral amyloid angiopathy (CAA). However, it is also possible that cerebrovascular disease could contribute to the presence of MBs in AD. Subjects with MBs are at a greater risk of bleeds which could impact the use of anti-coagulation treatment approaches.

The presence of CAA has been particularly associated with AD and studies have demonstrated that MBs occur in 12-33% of subjects with typical Alzheimer's dementia, with a large proportion of subjects showing multiple MBs. The presence of MBs has been associated with older age and a greater degree of white matter hyperintensities (WMH) in Alzheimer's dementia. The association between MBs and WMH, a marker of cerebrovascular disease, suggests cerebrovascular disease may also play a role in the etiology of MBs in AD. However, approximately 16% of AD subjects do not present with episodic memory loss, but instead display language problems such as poor naming and impaired sentence repetition, or visuospatial and visual perceptual deficits, and are referred to as atypical AD. Since AD is associated with CAA, one would assume that CAA and hence MBs, would also occur in atypical AD, although no studies have assessed MBs in atypical AD.

Amyloid-binding ligands, such as Pittsburgh Compound B (PiB), that can be detected using PET scanning have now been developed and provide an invaluable biomarker to infer the presence of β-amyloid. The presence of CAA has been shown to be associated with elevated PiB uptake, and hence the assessment of PiB-PET in subjects with MBs will provide important information on the association of MBs and β-amyloid deposition in AD.

The goal of the study is to assess the associations between MBs and demographic/clinical features, assess the associations between MBs and imaging features as well as a possible correlate to the number of MBs a subject has in atypical AD.

Patients found to be eligible and willing to enroll in this study will be asked to undergo a Neurologic Examination, Neuropsychometric testing, an MRI scan, and a PiB PET scan of the brain. This will be done over a period of two days at the Mayo Clinic in Rochester, Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 21
* will have an informant/study partner who will be able to provide independent evaluation of functioning
* must fulfill clinical diagnostic criteria for atypical AD, and hence should either have a chief complaint of difficulty with language and fulfill criteria for logopenic variant of primary progressive aphasia, or present with visuospatial/perceptual deficits and fulfill criteria for posterior cortical atrophy
* speaks English as their primary language (including bilingual patients whose primary language is English)
* agrees to and is eligible to undergo MRI and PET scanning
* if woman of child bearing age, must agree to pregnancy test no more than 48 hours before the PET scans

Exclusion Criteria:

* subjects with concurrent illnesses that could account for the presenting syndrome, such as traumatic brain injury, strokes or developmental syndromes
* subjects meeting criteria for another neurodegenerative disease, particularly typical Alzheimer's dementia
* women that are pregnant or post-partum and breast-feeding
* subjects will also be excluded if MRI is contraindicated (metal in head, cardiac pace maker, e.t.c.), if there is severe claustrophobia, and if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma or intracranial neoplasm)
* subjects will also be excluded if they do not have an informant, do not consent to research or do not complete all components of the study (neurological exam, neuropsychometric tests, MRI, PiB PET)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with and without microbleeds | up to day 2 of study

SECONDARY OUTCOMES:
Percentage of white matter hyperintensity burden on MRI and ratio of amyloid burden on PiB PET scan | Study entry, approximately day 1 or day 2 of study
Number of microbleeds per subject | Study entry, approximately day 1 or day 2 of study

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Whitwell, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States